CLINICAL TRIAL: NCT03857919
Title: Randomized, Controlled Trial to Evaluate the Safety and Effectiveness of the TearCare® System in the Treatment of the Signs and Symptoms of Dry Eye Disease
Brief Title: TearCare System to Treat Dry Eye Disease
Acronym: OLYMPIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sight Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06196
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-08

CONDITIONS: Dry Eye; Meibomian Gland Dysfunction
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TearCare (Experimental): Subjects will have heat applied to the eyelids for 15 minutes followed by manual expression of the meibomian glands.
  Interventions: Device: TearCare
- LipiFlow (Active Comparator): Subjects will have heat and pressure applied to the eyelids for 12 minutes.
  Interventions: Device: LipiFlow

INTERVENTIONS:
Device: TearCare — The TearCare SmartLids will be applied to the external surface of each eyelid. The TearCare System will be turned on and heat will be delivered to the eyelids for 15 minutes. Immediately following the thermal portion of the procedure, the SmartLids will be removed and the doctor will manually express the meibomian glands.
  Arms: TearCare
Device: LipiFlow — The LipiFlow activators will be placed between the inner eyelid and the corneal surface of each eye. The LipiFlow System will be turned on and heat and pressure will be delivered to each eyelid for 12 minutes.
  Other Names: Thermal Pulsation
  Arms: LipiFlow

SUMMARY:
In this study, the TearCare System will be compared with the LipiFlow Thermal Pulsation System in patients with dry eye disease. The objective is to demonstrate that the TearCare System is safe and effective in relieving the signs and symptoms of dry eye disease.

DETAILED DESCRIPTION:
The primary objective of this study was to demonstrate the safety and effectiveness of a single TearCare System treatment compared to a single LipiFlow treatment in relieving the signs and symptoms of dry eye disease. This study was conducted to collect data to support a modification to the TearCare indication for use to read as follows, "The TearCare® System is indicated for the treatment of the signs and symptoms of dry eye disease (DED)."

ELIGIBILITY:
Key Inclusion Criteria:

* At least 22 years of age
* Reports dry eye symptoms within the past 3 months
* Reports having to use artificial tears or lubricants regularly over the past month to relieve dry eye symptoms.
* OSDI Score of 23-79
* TBUT of ≤7 seconds in both eyes
* Meibomian gland obstruction in both eyes based on a total Meibomian Gland Secretion Score ≤12 in each eye.
* At least 15 glands in each lower eyelid should be expressible, with a sterile cotton swab, at the slit lamp.
* Best corrected visual acuity of 20/100 or better in both eyes.
* Willing and able to comply with the study procedures and follow-up
* Willing and able to provide informed consent
* English-speaking

Key Exclusion Criteria:

* Use of any of the following medications:

  1. Restasis or Xiidra within 60 days prior to enrollment;
  2. Antihistamines (oral or topical) within 10 days prior to enrollment;
  3. Systemic medication(s) (other than anti-histamines) that is known to cause ocular dryness (e.g. diuretics, anti-hypertensives, anti-depressants, hormone therapy) and whose dose of this medication(s) has not been stable within 30 days prior to enrollment. There must be no anticipated adjustments to the dose of these medications for the duration of the trial;
  4. Accutane (at any time);
  5. Oral tetracyclines or azithromycin within 30 days prior to enrollment; or
  6. Topical ophthalmic antibiotics, anti-glaucoma medications, steroids, non-steroidal anti-inflammatory medications within 30 days prior to enrollment.

     NOTE: Use of any of the above medications (with the exception of 1c) is not permitted during the 1 month follow-up period.
* Any of the following dry eye treatments:

  1. Office-based dry eye treatment (e.g. IPL, thermal pulsation [Lipiflow], etc.) within 12 months prior to enrollment;
  2. Meibomian gland expression within 6 months prior to enrollment;
  3. Blephex or debridement within 3 months prior to enrollment is an exclusion;
  4. Punctal occlusion or punctal plug placement within 30 days prior to enrollment;
  5. Use of TrueTear device within the past 2 weeks. (Subjects must refrain from using the TrueTear device for the duration of the study.); or
  6. Any history of meibomian gland probing
* History of eyelid, conjunctiva or corneal surgery (including refractive surgery) within the past year. In addition, subjects with any history of the following are excluded: chalazion surgery, surgery on the tarsal conjunctiva, radial keratotomy (RK), complicated blepharoplasty, lid reconstruction, or significant complications post-refractive surgery.
* Contact lens use within the past 2 weeks. (Subjects must refrain from wearing contact lenses during the 1-month follow-up.)
* History of Ocular Herpes Simplex or Ocular Herpes Zoster
* Any active, clinically significant ocular or peri-ocular infection or inflammation
* Recurrent clinically significant eye inflammation, other than dry eye, within 3 months prior to enrollment
* Clinically significant anterior blepharitis. In addition, collarettes or flakes of more than one quarter of the eyelid are excluded.
* Clinically significant eyelid abnormalities in either eye (e.g. entropion/ectropion, blepharospasm, aponeurotic ptosis, lagophthalmos, distichiasis, trichiasis).
* Clinically significant dermatologic or cutaneous disease of the eyelid or periocular area.
* In the clinical judgement of the investigator, meibomian glands have significant capping, atrophy, or are unable to be expressed, digitally or with a sterile cotton swab.
* Clinically significant ocular surface abnormalities that may affect tear film distribution or treatment (e.g. pterygium, anterior membrane dystrophy, Salzmann's nodules, etc.)
* Corneal surface abnormalities such as corneal epithelial defects (other than punctate staining), ulcers, corneal epithelial dystrophies, keratoconus, and ectatic disease of the cornea
* Any active, clinically significant allergic, vernal, or giant papillary conjunctivitis.
* Ocular trauma within 3 months prior to enrollment.
* Known history of diminished or abnormal facial, periocular, ocular or corneal sensation
* Systemic diseases resulting in dry eye (e.g. autoimmune diseases such as Sjogren's syndrome, rheumatoid arthritis, lupus, Graves' disease, sarcoidosis, etc.)
* Subject is currently using Retin A or Latisse.
* Subject has permanent eyeliner/lid tattoos, eyelash extensions or wears false eyelashes.
* Subject is currently using Lash Boost.
* Allergies to silicone tissue adhesives
* Participation in another ophthalmic clinical trial within one year prior to enrollment. Subject must also be willing to refrain from another ophthalmic study for the duration of the study.
* Co-existing condition, either ocular or non-ocular that, in the judgement of the investigator could affect the safety or effectiveness of treatment or the compliance of the subject to the protocol. For example, subjects who are pregnant or nursing or have active, wet macular degeneration are excluded.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Dickerson, PhD, Study Director — Sight Sciences
Locations (10):
- United States (10):
  - Schwartz Laser Eye Center, Scottsdale, Arizona
  - Harvard Eye Associates, Laguna Hills, California
  - Eye Research Foundation, Newport Beach, California
  - Loh Ophthalmology Associates, Miami, Florida
  - Jackson Eye, Lake Villa, Illinois
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Kentucky Eye Institute, Lexington, Kentucky
  - Ophthalmology Associates, St Louis, Missouri
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Parkhurst NuVision, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holland EJ, Loh J, Bloomenstein M, Thompson V, Wirta D, Dhamdhere K. A Comparison of TearCare and Lipiflow Systems in Reducing Dry Eye Disease Symptoms Associated with Meibomian Gland Disease. Clin Ophthalmol. 2022 Aug 30;16:2861-2871. doi: 10.2147/OPTH.S368319. eCollection 2022. PMID 36065356

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TearCare | LipiFlow
Started | 115 | 120
Completed | 115 | 120
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TearCare | LipiFlow | Total
Number analyzed (Participants) | 115 | 120 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (14.0) | 55 (14.5) | 55.9 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 83 | 169
  Male | 29 | 37 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 19 | 40
  Not Hispanic or Latino | 94 | 101 | 195
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 104 | 109 | 213
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Tear Break Up Time [Mean (Standard Deviation); unit: seconds] — The TBUT was evaluated by measuring the time to breakup of the tear film following a complete blink when viewed through the slit-lamp using a cobalt blue filter. The TBUT was recorded using a stopwatch for each eye as the average of 3 measurements at each visit.
  seconds | 4.5 (1.2) | 4.5 (1.2) | 4.5 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Tear Break-Up Time (TBUT) From Baseline
Description: Tear Break-Up Time is the time measured to the first observation of a break in the tear film
Time Frame: 1 month
Population: Primary Analysis Population
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | TearCare | LipiFlow
Number analyzed (Participants) | 67 | 68
Seconds | 3.02 (4.41) | 2.58 (3.28)

2. Primary Outcome: Change in Meibomian Gland Secretion Score From Baseline
Description: The Meibomian Gland Secretion Score grades the consistency of secretions from the meibomian glands. Fifteen meibomian glands in each of the lower eyelids were gently pressed and the secretions were scored on the scale below. Sum of the grade (0 - 3) for each of the 15 glands. Range for this score is 0-45. A higher number indicates more normal meibomian gland activity.
  Score Description of Secretion:
  0 - Nothing
  1. - Toothpaste
  2. - Cloudy
  3. - Clear
Time Frame: 1 month
Population: Primary Analysis Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TearCare | LipiFlow
Number analyzed (Participants) | 67 | 68
score on a scale | 11.20 (11.13) | 11.09 (10.41)

3. Secondary Outcome: Mean Change in Ocular Surface Disease Index (OSDI) Score From Baseline
Description: The Ocular Surface Disease Index (OSDI) questionnaire is a validated questionnaire that consists of 12 questions to assess ocular symptoms, their impact on patient vision-related functioning, and environmental factors triggering the symptoms. Scale range is zero (best possible score) to 100 (worst possible score). Mean change is the average of the difference between Month 1 and baseline for each subject. A negative result represents improvement.
  OSDI Scale Dry Eye Grade 12 or less - Normal 13-22 - Mild 23-32 - Moderate 33 or greater - Severe
Time Frame: 1 month
Population: Primary Analysis Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TearCare | LipiFlow
Number analyzed (Participants) | 67 | 68
score on a scale | -27.88 (20.48) | -23.40 (17.71)

4. Secondary Outcome: Change in Corneal Staining Score From Baseline
Description: The structural effect of dry eye disease (DED) on subjects' ocular surface and its severity was assessed using corneal and conjunctival staining. The degree of staining was quantified using the NEI/Industry Grading System which scores 5 regions of the cornea and 6 regions of the conjunctiva using a scale from 0 to 3. On this scale, 0 indicates no staining and 3 indicates severe staining. The score for the regions of the cornea were added to obtain a total score that ranged from 0-15 where 0 indicates no ocular surface damage or dry eye.
Time Frame: 1 month
Population: Primary Analysis Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TearCare | LipiFlow
Number analyzed (Participants) | 67 | 68
score on a scale | -0.25 (1.98) | -0.57 (2.01)

5. Secondary Outcome: Change in Conjunctival Staining Score From Baseline
Description: The structural effect of dry eye disease (DED) on subjects' ocular surface and its severity was assessed using corneal and conjunctival staining. The degree of staining was quantified using the NEI/Industry Grading System which scores 5 regions of the cornea and 6 regions of the conjunctiva using a scale from 0 to 3. On this scale, 0 indicates no staining and 3 indicates severe staining. The score for the regions of the conjunctiva were added to obtain a total score that ranged from 0-18, where 0 indicates no ocular surface damage or dry eye.
Time Frame: 1 month
Population: Primary Analysis Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TearCare | LipiFlow
Number analyzed (Participants) | 67 | 68
score on a scale | -0.66 (2.26) | -0.78 (3.18)

6. Secondary Outcome: Change in Symptom Assessment in Dry Eye (SANDE) Scores From Baseline
Description: The SANDE instrument is a simple 2-item questionnaire, that focuses on the frequency and the severity of dry eye symptoms with each measured along a visual analog scale. SANDE, because of its simplicity, is often used in routine clinical practice. For the core questions, the frequency and severity scores are multiplied together, and the square root is taken to produce an overall SANDE score from 0 (best possible) to 100 (worst possible). The mean change from baseline to month 1 is the difference in the two scores. A negative result indicates improvement.
Time Frame: 1 month
Population: Primary Analysis Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TearCare | LipiFlow
Number analyzed (Participants) | 67 | 68
score on a scale | -38.21 (31.05) | -39.41 (25.97)

7. Secondary Outcome: Change in Eye Dryness Score (EDS) From Baseline
Description: Severity of dry eye symptoms assessed on a 100 mm visual analog scale (VAS) ranging from 'Never/Very comfortable' to 'All the time/Very severe' and scored from 0 to 100: "0" = no discomfort/very comfortable, "100" = very severe.
Time Frame: 1 month
Population: Primary Analysis Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TearCare | LipiFlow
Number analyzed (Participants) | 67 | 68
score on a scale | -35.43 (34.11) | -34.87 (26.99)

8. Secondary Outcome: Change in Total Number of Meibomian Glands Yielding Clear Liquid From Baseline
Description: This is a count of the number of glands scored as having clear secretions. Fifteen glands are scored. Total score ranges from 0-15 with 15 being the best.
Time Frame: 1 month
Population: Primary Analysis Population
Measure: Mean (Standard Deviation); unit: Number of meibomian glands
Arm/Group | TearCare | LipiFlow
Number analyzed (Participants) | 67 | 68
Number of meibomian glands | 1.82 (3.74) | 1.83 (3.54)

9. Secondary Outcome: Change in Total Number of Meibomian Glands Yielding Any Liquid From Baseline
Description: This is a count of the number of glands scored as having any secretions. Fifteen glands are scored. Total score ranges from 0-15 with 15 being the best.
Time Frame: 1 month
Population: Primary Analysis Population
Measure: Mean (Standard Deviation); unit: Number of meibomian glands
Arm/Group | TearCare | LipiFlow
Number analyzed (Participants) | 67 | 68
Number of meibomian glands | 4.31 (3.66) | 4.35 (3.42)

ADVERSE EVENTS:
Time Frame: 1 Month
Arm/Group | TearCare | LipiFlow
All-Cause Mortality (participants affected / at risk) | 7/115 | 8/120
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/120
Other Adverse Events (participants affected / at risk) | 7/115 | 8/120
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TearCare (N=115) | LipiFlow (N=120)
Chalazion (Eye disorders) | 1 (1) | 0 (0)
Superficial Punctate Keratitis (SPK) (Eye disorders) | 1 (1) | 0 (0)
Decrease in BCVA (Eye disorders) | 2 (2) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 1 (1)
Conjunctival Injection (Eye disorders) | 1 (1) | 0 (0)
Iritis (Eye disorders) | 1 (1) | 0 (0)
Epiphora (Eye disorders) | 0 (0) | 1 (1)
Foreign Body Sensation (Eye disorders) | 0 (0) | 2 (2)
Ocular Pain (Eye disorders) | 0 (0) | 1 (1)
Corneal Abrasion (Eye disorders) | 0 (0) | 1 (1)
Dry Eye Disease (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/19/NCT03857919/Prot_SAP_001.pdf